CLINICAL TRIAL: NCT01717144
Title: EVALUATION OF A THERAPEUTIC EDUCATION PROGRAMME IN PARKINSON'S DISEASE
Brief Title: Education in Therapy of Parkinson's Disease
Acronym: ETPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08 150 07
Record Dates: First submitted 2012-10-22; First posted 2012-10-30 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Parkinson Disease
Keywords: therapeutic education; Parkinson's disease; quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- traditional medical care (No Intervention): patients benefiting of a traditional medical care
- therapeutic education program (Experimental): The educational program consisted of both individual and collective educational consultations with a therapeutic education nurse
  Interventions: Behavioral: therapeutic education program

INTERVENTIONS:
Behavioral: therapeutic education program — The educational program consisted of both individual and collective educational consultations with a therapeutic education nurse
  Arms: therapeutic education program

SUMMARY:
Parkinson's disease (PD) has considerable impact on motor, psychological and social activities and significantly affects the quality of life of patients and their families. To improve the medical care of PD patients, the investigator have developed an educational program specific to PD.

The principal aim of this study is to evaluate the therapeutic education Program, comparing the quality of life of PD patients with or without the educational program after six month and one year follow-up.

The secondary aims are to evaluate the evolution of motor and psychological states in these 2 groups of patients and to compare the medical costs.

This is a monocentric, comparative, prospective randomised study. The investigators will evaluate 120 PD patients, 60 patients benefiting of the educational program and 60 patients with a traditional medical care. Quality of life of PD patients is evaluated using a specific scale (PDQ39) and a generalist scale (SF36) at 6 and 12 months. Motor and psychological states were assessed with UPDRS and HAD Scales. The educational program consisted of both individual and collective educational consultations.

The investigators supposed that the therapeutic education program will improve the quality of life of PD patients. The supposition that this improvement will correlate with the motor and psychological states.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of Parkinson's disease according to the criteria of the UKPDSBB
* Parkinson's disease patients with a score ≤4 on the Hoehn and Year scale
* Patient without cognitive disorders
* Patients treated with dopaminergic antiparkisonian drugs (L-DOPA, dopamine agonists,ICOMT…) or DBS stimulation (since at least 3 month)
* Patients able to fulfil self-administered questionnaire
* Patients affiliated to a social protection program

Exclusion Criteria:

* - Patients suffering from an other pathology causing chronic pain (rheumatic disease, traumatic or orthopaedic pathologies…)
* Parkinson's disease patients with a score>5 on the Hoehn and Yahr scale
* Patients suffering of parkinsonism induce by drugs
* Patients with important tremors during a OFF conditions
* Patients ever included in another study
* Patients with severe psychiatric disease
* Patients under tutelage, curatelle or law protection
* Patients included in an other clinical study
* Patients unable to fulfil scales of the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Quality of life with the PDQ39 scale | 1 year

SECONDARY OUTCOMES:
Quality of life with the SF36 scale | 1 year
the motor state with UPDRS (Unified Pakinson's disease Rating Scale) | 1 year
The psychological state with HAD (Hospital Anxiety and Depression) scale | 1 year
Evaluation of social adaptation with SAS-SR (Social adjustement Scale Sel-Report) scale | 1 year
Evaluation of medical costs | over the 12 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- UH Toulouse, Toulouse, France

REFERENCES:
- [Result] Ory Magne F, Arcari C, Canivet C, Sarrail M, Fabre MH, Mohara C, Brefel Courbon C. [A therapeutic educational program in Parkinson's disease: ETPARK]. Rev Neurol (Paris). 2014 Feb;170(2):128-33. doi: 10.1016/j.neurol.2013.08.007. Epub 2013 Nov 20. French. PMID 24267951